CLINICAL TRIAL: NCT01026389
Title: Efficacy Evaluation of Dotarem®-Enhanced MRA Compared to Gadovist®-Enhanced MRA in the Diagnosis of Clinically Significant Abdominal or Limb Arterial Diseases
Brief Title: Efficacy Evaluation of Dotarem Compared to Gadovist in the Diagnosis of Peripheral Arterial Disease
Acronym: DALIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DGD 44-045
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Peripheral Arterial Disease
Keywords: MRA-Contrast agent comparison in peripheral disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — gadoterate meglumine; gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; gadobutrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gadovist (Active Comparator): Patient received contrast-enhanced MRA with Gadovist
  Interventions: Drug: Gadovist
- Dotarem, interventional (Experimental): Patients received contrast-enhanced MRA with Dotarem
  Interventions: Drug: Dotarem

INTERVENTIONS:
Drug: Dotarem — DOTAREM, 0.1 mmoL/kg (0.2 mL/kg), intravenous (I.V.) bolus
  Other Names: gadoterate; Gd-Dota
  Arms: Dotarem, interventional
Drug: Gadovist — Gadovist, 0.1mmol/kg (0.1mL/kg), intravenous (I.V.) bolus
  Other Names: gadobutrol
  Arms: Gadovist

SUMMARY:
This study is an efficacy evaluation of Dotarem®-enhanced magnetic resonance angiography (MRA) compared to Gadovist®-enhanced MRA in the diagnosis of clinically significant abdominal or lower limb arterial diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years.
* Patient with infrarenal aorta or chronic lower limb ischemia with various clinical signs of gravity (stages II-IV according to the classification of Leriche and Fontaine) or/and Doppler ultrasonography indicating abdominal or lower limb arteriopathy.
* Patient scheduled for a conventional X-Ray angiography (intra-arterial Digital Substraction Angiography = DSA) within 30 days of MRA with a minimum time interval of at least 24 hours between the 2 examinations.

Exclusion Criteria:

* Patient planned to undergo therapeutic intervention in abdominal or lower limb vessels between the time of MRA and X-ray Angiography will be performed.
* Patient who had a major cardiovascular event within 30 days prior to the inclusion.
* Patient treated with unilateral hip replacement, abdominal aortic or iliac graft or stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AKH hospital, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period between october 2009 and January 2011. Patients were recruited in hospitals.
Pre-assignment Details: 3 patients were not randomized: 2 patients because of technical issue and one patient because of sponsor decision (inclusion period finished/ number of evaluable patients achieved)
Groups:
- Dotarem: Patients received contrast-enhanced MRA with Dotarem
Period: Overall Study
Arm/Group | Gadovist | Dotarem
Started | 93 | 93
Completed | 88 | 88
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 3
Not completed — change of treatment, patient moved | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gadovist | Dotarem, Interventional | Total
Number analyzed (Participants) | 93 | 93 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 48 | 96
  >=65 years | 45 | 45 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 66.5 (10.2) | 66.8 (10.6) | 66.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 72 | 75 | 147
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 18 | 37
  France | 16 | 20 | 36
  Germany | 7 | 7 | 14
  Italy | 16 | 16 | 32
  Spain | 35 | 32 | 67

OUTCOME MEASURES:

1. Primary Outcome: Intra-patient Accuracy (Percent Agreement), On-site Data
Description: intra-patient accuracy (percent agreement) of each type of MRA examination (Dotarem® or Gadovist®-enhanced MRA) in assessing the lesions of the concerned territory as compared with the gold standard, X-ray angiography.
Time Frame: up to one month
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of agreement
Arm/Group | Gadovist | Dotarem, Interventional
Number analyzed (Participants) | 87 | 86
percentage of agreement | 77.1 (19.6) | 80.6 (16.1)

2. Secondary Outcome: Intra-patient Accuracy, in Off-site Readings
Description: • Intra-patient accuracy (percent agreement) of each type of MRA examination (Dotarem® or Gadovist®-enhanced MRA) in assessing the lesions of the concerned territory as compared with the gold standard, X-ray angiography, in off-site readings, using the same methodology as that used for the primary criterion
Time Frame: up to one month
Population: Ecah images from each patient were analysed by two external readers, this means that each patient was analyzed twice.
  Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of agreement
Units Other Than Participants: images
Arm/Group | Gadovist | Dotarem, Interventional
Number analyzed (Participants) | 78 | 76
Number analyzed (images) | 156 | 152
percentage of agreement | 75.1 (15.3) | 73.9 (16.7)

3. Secondary Outcome: Specificity
Description: Specificity of Dotarem® and Gadovist®-enhanced MRA examinations at the segment and the patient levels (gold standard = x-ray angiography) in on-site readings; no stenosis and non significant stenosis were grouped as one class (non significant stenosis = negative segment).
Time Frame: up to one month
Population: per protocol population
Measure: Number; unit: negative segments in MRA
Units Other Than Participants: Negative segment with gold standard
Arm/Group | Gadovist | Dotarem, Interventional
Number analyzed (Participants) | 79 | 77
Number analyzed (Negative segment with gold standard) | 819 | 824
negative segments in MRA | 756 | 763

4. Secondary Outcome: Sensitivity
Description: sensitivity of Dotarem® and Gadovist®-enhanced MRA examinations at the segment and the patient levels (gold standard = x-ray angiography) in on-site; moderate, severe stenosis and occlusion were grouped as one class (significant stenosis = positive segment).
Time Frame: up to one month
Population: Per protocol population
Measure: Number; unit: positive segment with MRA
Units Other Than Participants: positive segment with gold standard
Arm/Group | Gadovist | Dotarem, Interventional
Number analyzed (Participants) | 79 | 77
Number analyzed (positive segment with gold standard) | 238 | 264
positive segment with MRA | 168 | 191

ADVERSE EVENTS:
Time Frame: 15 months in total For each patient, adverse events were collected from signature of inform consent form to the end of the DSA
Arm/Group | Gadovist | Dotarem, Interventional
Serious Adverse Events (participants affected / at risk) | 0/93 | 1/93
Other Adverse Events (participants affected / at risk) | 2/92 | 2/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadovist (N=93) | Dotarem, Interventional (N=93)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) — Not related, occured prior to administration of study treatment
carotid stenosis (Nervous system disorders) | 0 (0) | 1 (1) — Not related, occured prior to administration of study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gadovist (N=92) | Dotarem, Interventional (N=92)
Folliculis (Infections and infestations) | 0 (0) | 1 (1) — Not related, mild
contrast extravasation (General disorders) | 1 (1) | 0 (0) — Not related, mild
burning (Nervous system disorders) | 0 (0) | 1 (1) — Possibly related, mild
heat sensation in the face (Vascular disorders) | 1 (1) | 0 (0) — Possibly related, mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less